CLINICAL TRIAL: NCT07045389
Title: Influence of the Sinus Floor-to-lower Window Margin Distance on Outcomes of Bone Window Repositioning in Lateral Sinus Floor Elevation With Simultaneous Implant Placement: A Retrospective Study
Brief Title: Influence of the Sinus Floor-to-lower Window Margin Distance on Outcomes of Bone Window Repositioning in Lateral Sinus Floor Elevation With Simultaneous Implant Placement
Status: Completed | Type: Observational
Sponsor: Guoli Yang (Other)
Collaborators: National Natural Science Foundation of China (Other Government); The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Guoli Yang, Professor, The Dental Hospital of Zhejiang University School of Medicine
Organization: The Dental Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: 2024-204R; 82271001; 82370991; 2022KY872 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC); Zhejiang Provincial Department of Science and Technology)
Record Dates: First submitted 2025-06-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Sinus Floor Elevation
Keywords: clinical research; cone-beam computed tomography; sinus floor elevation; bone window repositioning; sinus floor-to-lower window margin distance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DSLW ≥ 3 mm: Patients undergoing lateral sinus floor elevation with simultaneous implant placement, in whom the distance from the sinus floor to the lower edge of the lateral window is greater than or equal to 3 mm.
- DSLW < 3 mm: Patients undergoing lateral sinus floor elevation with simultaneous implant placement, in whom the distance from the sinus floor to the lower edge of the lateral window is less than 3 mm.

SUMMARY:
The goal of this observational study is to evaluate how the vertical distance from the sinus floor to the lower margin of the lateral window affects bone regeneration and implant outcomes after lateral sinus floor elevation with simultaneous implant placement. The main question it aims to answer is:

Does a sinus floor-to-window margin distance ≥3 mm lead to better bone augmentation and implant stability compared to a distance <3 mm?

This is a retrospective, single-center cohort study. Participants included patients who had previously undergone lateral sinus floor elevation with implant placement and had at least 6 months of postoperative follow-up. Cone-beam CT images were used to measure radiographic outcomes such as alveolar bone height and augmented volume.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Received lateral sinus floor elevation with bone window repositioning and simultaneous implant placement (LSFE with BWR and SIP) between 2019 and 2024
* No contraindications to implantation
* Complete medical and radiographic records available

Exclusion Criteria:

* Uncontrolled systemic diseases
* Incomplete medical or surgical records
* Missing preoperative or postoperative imaging data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lateral sinus floor elevation with simultaneous implant placement at a single academic hospital in China. Inclusion was based on availability of preoperative CBCT and a follow-up period of at least 6 months. Patients were grouped according to the vertical distance from the sinus floor to the lower margin of the lateral window.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
ABH at T1, ABH at T2, ABH change from T1 to T2, ESBG at T1, ESBG at T2, ESBG change from T1 to T2, BBH at T1, BBH at T2, BBH change from T1 to T2, PBH at T1, PBH at T2, PBH change from T1 to T2, AV at T1, AV at T2, AV change from T1 to T2 | T1 (immediately after surgery) and T2 (6 months after surgery)
  ABH at T1 (mm): Alveolar bone height measured immediately after surgery; ABH at T2 (mm): ABH measured 6 months after surgery; ABH change from T1 to T2 (%): ABH Calculated as ((T2 - T1) / T1) × 100%; ESBG at T1 (mm): Elevated sinus bone gain measured immediately after surgery; ESBG at T2 (mm): ESBG measured 6 months after surgery; ESBG change from T1 to T2 (%): ESBG Calculated as ((T2 - T1) / T1) × 100%; BBH at T1 (mm): Buccal bone height measured immediately after surgery; BBH at T2 (mm): BBH measured 6 months after surgery; BBH change from T1 to T2 (%): BBH Calculated as ((T2 - T1) / T1) × 100%; PBH at T1 (mm): Palatal bone height measured immediately after surgery; PBH at T2 (mm): PBH measured 6 months after surgery; PBH change from T1 to T2 (%): PBH Calculated as ((T2 - T1) / T1) × 100%; AV at T1 (mm³): Augmented volume measured immediately after surgery; AV at T1(mm³): AV measured 6 months after surgery; AV change from T1 to T2 (%): AV Calculated as ((T2 - T1) / T1) × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital, School of Stomatology, Zhejiang University., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the retrospective nature of the study and ethical considerations related to patient privacy.